CLINICAL TRIAL: NCT01258426
Title: Human Selenoprotein P Concentration With Glucose Tolerance Status
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Other Study IDs: SEPP1(DM)
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: SEPP1 Levels in Differnet Glucose Tolerance Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal, IGT, T2DM

SUMMARY:
Recently, seslenium(Se) has known as important regulator in metabolic status, lipid profile, atherosclerosis progression. SEPP1(selenoprotein P1)is a secreted protein from mainly liver. This protein is used as an index of selenium nutritional status. The association between the concentration of SEPP1(selenoprotein P1) in normal glucose tolerance,impaired glucose tolerance, type 2 diabetes is still a matter of debate. This cross sectional study will evaluate whether glucose status is matter in SEPP1 level.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 years old
* Not severe medical condition

Exclusion Criteria:

* metformin, insulin using type 2 diabetes

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total 180 patients Normal 60-IGT 60-T2DM 60
Sampling Method: Non-Probability Sample